CLINICAL TRIAL: NCT01980394
Title: Esophageal Stump Washout Reduces Free Intraluminal Tumor Cells During Resection of Carcinomas of the Esophagus and Cardia
Brief Title: Esophageal Stump Washout
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Liestal (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Liestal-2012-OES
Record Dates: First submitted 2013-08-30; First posted 2013-11-11 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Esophageal Cancer; Gastrooesophageal Cancer
Keywords: esophagus; gastro-esophegeal junction; cancer; tumor seeding; free viable tumor cells; surgery; intraluminal tumor cells; stump washout
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- prospective cohort study (Other)
  Interventions: Procedure: Esophageal Stump Washout

INTERVENTIONS:
Procedure: Esophageal Stump Washout — a washout of the closed esophageal stump with Ringer-solution (10 times 30ml) is performed by means of a transorally inserted 24F-Foley catheter. The first, fifth and tenth portion of the lavage fluid are collected and sent to cytological examination

SUMMARY:
Intraluminally shed viable tumor cells might contribute to local recurrence in cancer of the esophagus and the cardia. The aim of the the study was to establish a method of mechanical lavage of the remaining part of the esophagus and, hence, to reduce the intraluminal cancer cells before doing the esophageal anastomosis.

DETAILED DESCRIPTION:
See study protocol!

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cancer of gastro-esophageal junction with indication for surgery

Exclusion Criteria:

* missing informed consent

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Presence of intraluminal tumor cells in the remaining oesophageal stump | during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Christoph A. Maurer, Professor, Chairman of Surgery, Study Chair — Hospital of Liestal, Liestal, Switzerland
Locations (1):
- Kantonsspital Baselland, Liestal, Liestal, Basel-Landschaft, Switzerland